CLINICAL TRIAL: NCT00382356
Title: A Pilot Investigation of Dutasteride (Avodart) After Failure of Finasteride (Proscar) In the Management of Symptomatic Prostatic Enlargement/Hypertrophy (BPE/H)
Brief Title: Dutasteride After Failure of Finasteride In the Management of Symptomatic Prostatic Enlargement/Hypertrophy (BPE/H)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: North Florida/South Georgia Veterans Health System (Other)
Responsible Party: Principal Investigator, Unyime O. Nseyo, MD, PHYSICIAN, North Florida/South Georgia Veterans Health System
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AVODART-550-04
Record Dates: First submitted 2006-09-28; First posted 2006-09-29 (Estimated); Last update posted 2012-10-19 (Estimated); Status verified 2012-10

CONDITIONS: Benign Prostatic Hypertrophy
Keywords: Benign Prostatic Enlargement; Benign Prostatic Hypertrophy; Dutasteride; 5-alpha reductase inhibitors; Hormonal therapy
MeSH Terms: conditions — Prostatic Hyperplasia | interventions — Dutasteride

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- study drug (Experimental): Open label, single arm
  Interventions: Drug: Dutasteride

INTERVENTIONS:
Drug: Dutasteride — once daily dosing of 0.5mg Dutasteride for 12 months
  Other Names: Avodart

SUMMARY:
The study is to determine the safety and efficacy of Dutasteride in patients who have failed Finasteride therapy for their symptomatic benign prostatic enlargement/ hypertrophy (BPE/H).

DETAILED DESCRIPTION:
STUDY SUMMARY

TITLE: A Pilot Investigation of Dutasteride (Avodart) After Failure of Finasteride (Proscar) in the Management of Symptomatic Prostatic Enlargement/Hypertrophy OBJECTIVE: To determine the safety and efficacy of Dutasteride in patients who have failed Finasteride therapy for their symptomatic benign prostatic enlargement/ hypertrophy (BPE/H)

EXPERIMENTAL PLAN:

PATIENT SELECTION: Inclusion Criteria

1. Patients who demonstrate clinical evidence of failure after treatment with Finasteride for 12 or more months. Failure includes one or more of the following: (i) AUA SS > 10; (ii) Q-max < 10 cc/sec; (iii) Post void residual volume (PVR) >200cc.
2. Patients who remain subjectively symptomatic of LUTS secondary to BPH after treatment with Finasteride for at least six months.

Exclusion Criteria Patients with Neurogenic Bladder/LUTS secondary to neurologic disease Patients with the diagnosis of prostate cancer Patients with an allergy to Finasteride/Dutasteride

STUDY DESIGN AND DURATION:

This will be a single institution, open label pilot study involving 26 patients over 18-24 months. Each patient will be treated with the standard dose of Dutasteride for at least twelve months and followed for an additional 12 months.

EFFICACY AND SAFETY MEASUREMENTS:

Improvement in flowmetry, AUASS and PVR will be the primary outcome measures of efficacy. Quality of life measurement will be made also. The exploratory measures will include PSA and prostate volume. All adverse events including tolerability of the test agent will be recorded.

SUMMARY:

A positive result showing objective (AUASS, Q-max, PVR) and subjective (satisfaction index) improvement in these previously treated patients should engender interest in a multicenter study to confirm our data. The clinical import is that this population should be switched to Dutasteride without prolonged treatment with Finasteride for no additional benefit to the patient. A failure of treatment with one hormonal agent does not necessarily imply a lack of response to another agent of the same class.

ELIGIBILITY:
Inclusion Criteria:

1. Male with history of treatment with Finasteride for more than six months, and who demonstrate clinical evidence of failure (subjective symptoms of bladder outlet obstruction secondary to BPH-related LUTS; objective evidence: AUASS> 10;Q-max > 5cc/sec and <10c/sec (total voided volume of at least 125cc); post void volumes > 200cc)
2. Prostate volume > 30cc and < 80cc by transrectal ultrasound measurement
3. Total Serum PSA of < 15 ng/ml (corrected for Finasteride therapy)
4. Willingness and ability to give written informed consent and comply with study instructions and procedures.

Exclusion Criteria:

1. Clinical evidence of non-response to therapy with Finasteride for symptomatic BPH.
2. Total serum corrected PSA of greater than 15 ng/ml
3. History or clinical evidence of prostate cancer
4. History of acute urinary retention in three months prior.

Min Age: 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2004-11; Primary Completion 2009-07 (Actual); Study Completion 2009-07 (Actual)

PRIMARY OUTCOMES:
Urodynamic parameters (Qmax, Voided volume, and PVR) and AUASS | 12 months

SECONDARY OUTCOMES:
To assess safety and tolerability of Dutasteride | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Unyime O Nseyo, M.D., Principal Investigator — NF/SGVAHS